CLINICAL TRIAL: NCT03416439
Title: Effectiveness of a Lifestyle Intervention on Metabolic Syndrome. A Randomized Controlled Trial
Brief Title: Effectiveness of a Lifestyle Intervention on Metabolic Syndrome.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Simona Bo, Associate Professor, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AT2004
Record Dates: First submitted 2018-01-22; First posted 2018-01-31 (Actual); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Lifestyle Intervention

STUDY DESIGN:
Intervention Model Description: Lifestyle intervention program carried out by trained professionals versus standard, unstructured information given by the family physicians
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention arm (Experimental): lifestyle intervention program carried out by trained professionals
  Interventions: Other: lifestyle intervention
- control arm (No Intervention): standard, unstructured information given by the family physicians

INTERVENTIONS:
Other: lifestyle intervention — lifestyle intervention program carried out by trained professionals
  Arms: intervention arm

SUMMARY:
The investigators compared the effectiveness of a lifestyle intervention program carried out by trained professionals versus standard unstructured information on healthy lifestyle given by the family physicians in ameliorating the metabolic pattern of adults with multiple metabolic and inflammatory abnormalities.

DETAILED DESCRIPTION:
Intensive lifestyle intervention significantly reduces the progression to diabetes in high-risk individuals. It is unknown if a less intensive program might also be effective in the general population.

The investigators' aim was to compare the effectiveness of two different modalities that recommend a healthier lifestyle to reduce multiple metabolic abnormalities-a lifestyle intervention program with general recommendations carried out by trained professionals and standard unstructured information given by the family physician-in a dysmetabolic population-based cohort.

All subjects aged 45-64 (n=1,877) from 6 family physicians, representative of the local Health Districts of Asti (Northern Italy), were contacted. A metabolic screening was carried out on 1,658 subjects (88.3%) who accepted to participate.

Out of those subjects, 375 patients had either the metabolic syndrome (MS) or two components of the MS plus high-sensitivity C-reactive protein (CRP) serum values ≥3 mg/L, the cutoff point that differentiates high-risk groups for future cardiovascular events, and did not have any of the exclusion criteria.

Then,187 were randomly allocated to the intervention arm and 188 to the control arm; 18 and 22 individuals refused to participate, respectively. Finally, 169 patients were assigned to the lifestyle intervention program carried out by trained professionals (intervention arm) and 166 to the standard, unstructured information given by the family physicians (control arm). All participants received verbal, not-written, information, emphasizing the importance of a healthy lifestyle from their family physicians, who had previously participated in 3 meetings on standard practice lifestyle recommendations. No further individualized programs were offered to the control arm.

The intervention arm received detailed verbal and written individualized diet and exercise recommendations from trained professionals during five 60-min sessions covering diet, exercise, and behavior modifications (the first was a one-to-one meeting, the following were group sessions).

Anthropometric measurements and blood samples were collected from all participants at the beginning and at the trial end, after 1-year.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 45-64 from 6 family physicians, representative of the local Health Districts of Asti (Northern Italy)
* Presence of the metabolic syndrome (MS) or hs-CRP>3mg/l and 2 components of the MS

Exclusion Criteria:

* diabetes, cardiovascular diseases, chronic liver or kidney disease, advanced cancer

Ages: 45 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 335 (Actual)
Dates: Start 2004-09 (Actual); Primary Completion 2005-12 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Between-group change in the prevalence of the metabolic syndrome, defined by the National Cholesterol Education Program criteria | 1 year after randomization
  Metabolic syndrome was defined by the National Cholesterol Education Program criteria as the presence of ≥3 of the following five criteria: fasting glucose ≥6.1 mmol/L; blood pressure ≥ 130/85 mmHg; triglycerides ≥1.69 mmol/L; high-density lipoprotein (HDL) cholesterol <1.29 mmol/L (females) or <1.04 mmol/L (males), and waist circumference >88 cm (females) or >102 cm (males).

SECONDARY OUTCOMES:
Within- and between-group variations in arterial blood pressure | 1 year after randomization
Within- and between-group variations in weight values | 1 year after randomization
Within- and between-group variations in fasting glucose | 1-year after randomization
Within- and between-group variations in C-reactive protein values | 1-year after randomization
Within- and between-group variations in triglyceride values | 1-year after randomization
Within- and between-group variations in HDL-cholesterol values | 1-year after randomization